CLINICAL TRIAL: NCT00034697
Title: A Phase II Study of Temozolomide (SCH 52365) in Subjects With Brain Metastasis From Non-Small-Cell Lung Cancer
Brief Title: Study of Temozolomide in the Treatment of Brain Metastasis From Non-small-cell Lung Cancer (Study P02143)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02143; NCT00030836 (obsolete NCT alias)
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Metastases, Neoplasm; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms
Keywords: Brain mets; non-small cell lung cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
Brain metastases from solid tumors are diagnosed in more than 300,000 patients annually. Nonsmall cell lung cancer accounts for the majority of CNS mets. Treatment with whole brain radiation and steroids will improve neurologic symptoms in about 50% of patients although survival is short. This study will test the safety and efficacy of temozolomide in combination with radiation therapy in the treatment of patients with brain mets form nonsmall cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of non-small-cell lung cancer
* Stable systemic disease
* Maximum of one prior chemotherapy regimen for metastatic systemic disease
* Radiotherapy for local control or palliative bony lesions is allowed
* Karnofsky of greater than or equal to 70%
* Adequate hematologic, renal and liver function

Exclusion Criteria:

* Patients eligible for surgery of the brain
* Any previous chemotherapy for the brain metastasis
* Chemotherapy within 4 weeks or previous temozolomide
* Prior radiotherapy to the brain
* Radiation therapy to greater than 50% of the bone marrow
* Insufficient recovery from previous therapies
* Active nonmalignant systemic disease
* Inability to take oral medication
* Pregnant or nursing women
* Non use of adequate contraceptive techniques, negative urine pregnancy test is required
* Known AIDS related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-06-28 (Actual); Primary Completion 2003-01-30 (Actual); Study Completion 2003-01-30 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html